CLINICAL TRIAL: NCT06916117
Title: A Prospective Single Arm Trial of Neoadjuvant Chemo-immunotherapy Followed by Concurrent Chemoradiotherapy and Immunotherapy in Locally Advanced Cervical Cancer
Brief Title: Neoadjuvant Chemo-immunotherapy Followed by Concurrent Chemoradiotherapy and Immunotherapy in LACC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: immunotherapy-LACC
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: immunotherapy; LACC; chemoradiotherapy
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): Neoadjuvant chemotherapy (TP regimen) combined with PD-1 inhibitor was given, followed by concurrent chemoradiotherapy (cisplatin and PD-1 inhibitor) , and PD-1 inhibitor maintenance was given sequenced after RT.
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT)

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NACT) — Neoadjuvant chemotherapy:
  The neoadjuvant regimen prior to radiotherapy consists of paclitaxel 135-175 mg/m², cisplatin 75 mg/m², and Sintilimab 200 mg, administered every 3 weeks for 2 cycles.
  Concurrent chemoradiotherapy:
  Radical dose to the pelvic concurrent with cisplatin.
  Consolidative immunotherapy:
  Following the completion of chemoradiotherapy, Sintilimab consolidation therapy will be administered based on treatment efficacy and the patient's physical condition, for a total of 6 cycles, starting 3-4 weeks after chemoradiotherapy.

SUMMARY:
Concurrent chemoradiotherapy -immunotherapy followed by ICI maintenance was proved to improve the PFS by the Keynote-A18 in the LACC patients, and still more than 30% progressed. Neoadjuvant chemo-immunotherapy in LACC resulted in higher pCR rate. This prospective single arm study is to investigate the efficacy and safety of neoadjuvant immuno-chemotherapy followed by concurrent chemoradiotherapy and consolidative immunotherapy in LACC patients.

DETAILED DESCRIPTION:
This prospective single arm study aims to investigate the efficacy and safety of neoadjuvant immuno-chemotherapy followed by concurrent chemoradiotherapy and consolidative immunotherapy in LACC patients. Patients will be given two cycles of TP regimen + Sintilimab, followed by concurrent chemoraiotherapy, and consolidative 6 cycles of Sintilimab.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age between 18 and 75; (2)Untreated patients with pathologically proven squamous carcinoma; (3)T3-4N1-2M0 cervical cancer; (4)Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1; (5)Adequate hematological, renal and hepatic functions: (6)Hemoglobin > 8.0 g/dl ; Neutrophils > 2000 cells/μl; Leukocytes > 4 × 109/L; Platelets > 100 × 109/L; Serum urea nitrogen (BUN) ≤ 1.5 × upper normal limit (UNL); Serum creatinine (Cr) ≤ 1.5 × upper normal limit (UNL); Serum ALT/AST ≤ 2.5× UNL; Serum Total bilirubin ≤ 1.5× UNL; (7)Life expectancy > 6 months; (8)Eligible for concurrent chemoradiotherapy assessed by principle investigator; (9)No obvious active bleeding; (10)Written informed consent must be available before study registration.

Exclusion Criteria:

* (1)Recurrent or distant metastatic disease; (2)Prior malignancies (other than curable non-melanoma skin cancer) within 5 years; (3)Active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of substantial amount of hormones or other immunosuppressants; (4)Patients who need to receive systemic corticosteroids (dose equivalent to or higher than prednisone 10mg qd) or other immunosuppressants within 14 days before enrollment or during the study; (5)Vaccination of live attenuated vaccine 30 days before enrollment, or planned vaccination of live attenuated vaccine during the study; (6)Previous organ transplantation or HIV patients; (7)Allergic to macromolecular proteins /monoclonal antibodies, or to any test drug component; (8)Active acute or chronic viral hepatitis B or C. Hepatitis B virus (HBV) DNA> 2000 IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA> 10^3 copies/ml.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 30 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression disease free survival | 2 year
  the time interval from the date of treatment to disease progression, local or distant recurrence

SECONDARY OUTCOMES:
Adverse events | one year from the start of immunotherapy
  The number and incidence of adverse events and serious adverse events will be tabulated according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided